CLINICAL TRIAL: NCT01755871
Title: The Long-term Effect of Fingolimod on Circulating Immunocompetent Mononuclear Cells in Patients With Multiple Sclerosis
Brief Title: Long-term Effect of Fingolimod on Circulating Immunocompetent Mononuclear Cells in Patients With Multiple Sclerosis
Acronym: BiobankII
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: lack of recruitment
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FINGOHHU
Record Dates: First submitted 2012-12-19; First posted 2012-12-24 (Estimated); Last update posted 2016-06-09 (Estimated); Status verified 2015-06

CONDITIONS: Relapsing Remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Fingolimod Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fingolimod (Experimental): Gilenya 0,5mg per day, oral
  Interventions: Drug: Fingolimod

INTERVENTIONS:
Drug: Fingolimod — 0,5mg Fingolimod once a day
  Other Names: Gilenya

SUMMARY:
The purpose of this study is to explore immunomodulatory and immunosuppressive mechanisms of action of fingolimod in patients with Relapsing remitting multiple Sclerosis to collect data on biomarkers after initiation of fingolimod treatment.

DETAILED DESCRIPTION:
After treatment with fingolimod the blood of the patients will be collected at different time points to examine the changes of T cells, B cells and biomarkers.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent from patients capable of giving or withholding full informed consent must be obtained before any assessment is performed in this trial.
2. Male or female subjects aged 18-65 years.
3. Subjects with relapsing remitting forms of MS defined by 2010 revised McDonald criteria (see Appendix).
4. Patients with high disease activity despite treatment with a disease modifying therapy (≥ 1 relapse in the previous year, ≥ 9 hyperintense T2 lesions or ≥1 Gd-enhancing lesion or "non-responding" which could be defined as unchanged or increased relapse rate or ongoing severe relapses compared to previous year) or patients with rapidly evolving severe RRMS (e.g. ≥ 2 relapses with disease progression in one year and ≥ 1 Gd-enhancing lesion or with a significant increase in T2 lesions compared to a recent MRI).
5. Patients with Expanded Disability Status Scale (EDSS) score of 0-6.5 (see Appendix).
6. Sufficient ability to read, write, communicate and understand

Exclusion Criteria:

1. Patients with a manifestation of MS other than relapsing remitting MS.
2. Patients with a history of chronic disease of the immune system other than MS, which requires systemic immunosuppressive treatment, or a known immunodeficiency syndrome.
3. History or presence of malignancy (other than localized basal cell carcinoma of the skin and carcinoma in situ of the cervix) in the last 5 years
4. Diabetic patients with moderate or severe non-proliferative diabetic retinopathy or proliferative diabetic retinopathy and uncontrolled diabetic patients with HbA1c > 7%.
5. Diagnosis of macular edema during Baseline Visit (patients with a history of macular edema will be allowed to enter the study provided that they do not have macular edema at the ophthalmic baseline visit).
6. Patients with active systemic bacterial, viral or fungal infections, or known to have AIDS, Hepatitis B, Hepatitis C infection or to have positive HIV antibody, Hepatitis B surface antigen or Hepatitis C antibody tests.
7. Negative for varicella-zoster virus IgG antibodies at Baseline.
8. Have received any live or live attenuated vaccines (including for varicella-zoster virus or measles) within 1 month prior to baseline.
9. Patients who have received total lymphoid irradiation or bone marrow transplantation.
10. Patients who expect to be treated with any disease modifying drugs (DMD) during the study (i.e. IFN-β, glatiramer acetate); however no washout is needed for DMDs prior to baseline.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-01; Primary Completion 2016-01 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Reduction of CD4+ and CD8+ naïve T cells (CCR7+ CD45RA+) and central memory T cells (CCR7+CD45RA-), and an elevation of effector memory T cells (CCR7- CD45RA-) by examining the blood | Day 0, Day 28, Day 84, Day 168, Day 336, Day 504, Day 672 after treatment
  The primary endpoints are the reduction of CD4+ and CD8+ naïve T cells (CCR7+ CD45RA+) and central memory T cells (CCR7+CD45RA-), and an elevation of effector memory T cells (CCR7- CD45RA-)in the blood, and to study the effect of Fingolimod on Th17 cells by studying their signature cytokines (IL-17, IL-21, IL-22) as well as signature transcription factors (ROR-gamma-t, ROR-alpha, STAT3, Runx1) in peripheral venous blood over 2 years versus baseline.

SECONDARY OUTCOMES:
To investigate changes from baseline in B Lymphocytes, monocytes and NK cells in the blood after treatment with fingolimod | Day 0, Day 28, Day 84, Day 168, Day 336, Day 504, Day 672 after treatment
  To investigate changes from baseline in B Lymphocytes, monocytes and NK cells in the blood after treatment with fingolimod. This will be assessed by studying surface markers by FACS analysis for B lymphocytes (CD19, CD20, CD69), monocytes (CD14), NK cells (CD56).

OTHER OUTCOMES:
Change of the biomarkers BDNF, NGF, CNTF and LIF in the blood during treatment with fingolimod | Day 0, Day 28, Day 84, Day 168, Day 336, Day 504, Day 672 after treatment
  The exploratory endpoints are the change from baseline in the biomarkers BDNF, NGF, CNTF and LIF in the blood. The changes in mRNA expression and serum protein levels will be analysed in peripheral blood as a result of fingolimod treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Bernd Kieseier, Prof., Principal Investigator — Heinrich Heine Universität Düsseldorf
Locations (1):
- Heinrich Heine Universität Düsseldorf, Düsseldorf, Nord-Rhein Westfahlen, Germany